CLINICAL TRIAL: NCT05211999
Title: The Effect of Precede-Proceed Model Based Simulation Experience in Needlestick and Sharps Injuries Among Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Azize Karahan, Lecturer, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-19/26
Record Dates: First submitted 2021-12-19; First posted 2022-01-27 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Needlestick Injuries
Keywords: Needlestick Injuries; Healthcare workers; Simulation; Precede-process model; Model based learning
MeSH Terms: conditions — Needlestick Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Precede-Proceed Model Based Simulation Experience (Experimental)
  Interventions: Behavioral: Precede-Proceed Model Based Simulation Experience; Behavioral: Control Group
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Precede-Proceed Model Based Simulation Experience — The program was created on the basis of the PRECEDE-PROCEED Model.The program consists of eight phases. It will be carried out with theoretical training and simulation experience in the experimental group. In the control group, theoretical training will be given. Results will be followed.
  Arms: Precede-Proceed Model Based Simulation Experience
Behavioral: Control Group — No intervention in control group just theoretical education was done for them.
  Arms: Precede-Proceed Model Based Simulation Experience

SUMMARY:
Healthcare workers are exposed to many important risks that will negatively affect their health in their working environment. Among these risks, the most important threat is needlestick injuries. Needlestick injuries in healthcare workers with work-related injuries among studies, and the prevalence of injury remains high. In a study conducted by Gheshlagh et al. (2018), the prevalence of needlestick injuries in health workers was found to be 42.5%. It has been shown in studies conducted that the most common decision needlestick injuries among health workers are in nurses. In preventing injuries, preventing, and controlling negative behaviors related to the safe use of needlestick tools is among the most important strategies. In addition, the use of evidence obtained from interventional studies to prevent needlestick injuries in protection programs also plays an important role in prevention.

The importance of frequent and regular education about the subject has been mentioned especially in the studies conducted to prevent injuries. The World Health Organization (WHO) has published gold standards in the education of nurses and has recommended the use of electronic learning and simulation methods in the programs of nursing schools for learning and teaching according to these standards. It is important to use evidence-based practices to increase quality and competence by creating realistic clinical environments in nursing education. In this context, it is possible to use simulation-based experiences for educational purposes without exposure to infection control and employee safety in the clinical field.

In a study conducted by Nakamura et al. (2019), it was found that a simulation-based training program was effective in infection control. Due to the limited number of studies aimed at protecting the health of healthcare workers and controlling infection, more simulation-based studies are needed in this area. In addition, conducting model-based studies in developing behavior in health workers will also increase success. One of these models, the Precede-Process Model, is an important guide for users in assessing the social, epidemiological, behavioral, and environmental spheres of society for planning and evaluating programs. In summary, the aim of the study is to evaluate the effect of the Precede-Process Model-based simulation training program on preventing needlestick injuries in nurses who are the occupational group most exposed to injury.

ELIGIBILITY:
Inclusion Criteria:

* 0-1 years of experience in the profession,
* Nurses who volunteered to participate in the study,

Exclusion Criteria:

* Nurses who graduated from Acıbadem Mehmet Ali Aydınlar University
* Nurses who have worked in the profession for more than one year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Level | Immediately after the simulation
  The Student Satisfaction and Self-Confidence in Learning Scale: This instrument is a 13 item scale used to measure student satisfaction with the simulation activity (5 items) and self-confidence in learning(8 items). Responses are rated on a 5-point Likert scale with values ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher satisfaction and greater levels of self-confidence.
Simulation Design Features Level | Immediately after the simulation
  Simulation Design Scale: The Simulation Design Scale is a 20-item tool developed. Responses are rated on a 5 point Likert scale with the values ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate increased recognition of design features in simulation.
Recognition of Educational Best Practices in Simulation | Immediately after the simulation
  Education Practice Questionnaire: The instrument has 16 items and includes the following elements: learning (10 items); diverse ways of learning (2 items); high expectations (2 items); and collaboration (2 items). The instrument uses a 5-point Likert scale with categories ranging from 1 (strongly disagree with the statement) to 5 (strongly agree with the statement). Higher scores indicate increased recognition of educational best practices in simulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided